CLINICAL TRIAL: NCT05491135
Title: Hepatocytes Co-Encapsulated With Mesenchymal Stromal Cells in Alginate Microbeads for the Treatment of Acute Liver Failure in Paediatric Patients (HELP)
Brief Title: Hepatocyte Microbeads for Acute Liver Failure
Acronym: HELP
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: King's College Hospital NHS Trust (Other)
Collaborators: Medical Research Council (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 3571; 2019-000316-29 (EudraCT Number)
Record Dates: First submitted 2022-07-27; First posted 2022-08-08 (Actual); Last update posted 2022-08-08 (Actual); Status verified 2022-08

CONDITIONS: Acute Liver Failure
Keywords: Cell therapy; Paediatric Liver transplant
MeSH Terms: conditions — Liver Failure, Acute

STUDY DESIGN:
Intervention Model Description: ATIMP
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- HMB002 (Experimental): All patients will receive HMB002 infusion into the peritoneal cavity.
  Interventions: Biological: HMB002

INTERVENTIONS:
Biological: HMB002 — The solution containing microbeads will be infused manually into the peritoneal cavity under ultrasound guidance, with usually a 50ml syringe, as a single infusion or several infusions, to achieve in excess of 25 million hepatocytes per kilogram of the body weight.

SUMMARY:
Acute Liver Failure in children is associated with high mortality without liver transplantation. In addition, donor organ shortage makes it difficult to provide this treatment to every potential patient. Liver transplantation is life-saving but it carries the risk of major surgery and complications from lifelong anti-rejection drugs to suppress the immune system. If bridged across the immediate crisis following acute liver failure, the immense regenerative potential of the liver means that the patient's own liver may 're-grow'. This period is very time sensitive. Unfortunately, if the vital synthetic and detoxification function of the liver is not provided, the patient will often die before the liver can re-grow.

Transplantation of liver cells (hepatocytes) can provide this 'bridge' with considerable advantages over whole organ transplantation. Firstly, hepatocytes are derived from donor livers which are otherwise unsuitable for transplantation. Secondly, unlike whole organs, they can be frozen and stored, thus act as an 'off the shelf' treatment. Thirdly, the technique of hepatocyte transplantation within microbeads coated with alginate (a gel originating from seaweed) and infused into the abdominal cavity is much less invasive than liver transplantation. Finally, the alginate protects the cells against the body's immune system, avoiding the need for immunosuppressive drugs and the associated major risks. Furthermore, preclinical work in King's College Hospital has shown that the addition of support cells called mesenchymal stromal cells (MSCs), can significantly improve the ability of hepatocytes to survive and function within the alginate microbead.

The HELP trial is a Phase 1/2 safety and tolerability study of infusion of HMB002 (an optimal combination of hepatocytes and mesenchymal stromal cells put together in peptide-alginate microbeads) into paediatric patients with acute liver failure. This novel cellular therapy may act as a bridge treatment to liver transplant or lead to regeneration of the native liver.

DETAILED DESCRIPTION:
This is an open label, single centre study first in man study. The study will be conducted using the Simon two stage design. Nine patients will be recruited during stage 1 of the study. Once 9 patients have completed their 24 weeks visit, the study will stop for futility if only 2 or fewer patients have survived with the native liver. Otherwise, the study will progress to Stage 2 of recruitment, where the trial will continue to enroll a further 8 patients. A total of 17 patients will be recruited into the study (at the end of stages 1 and 2). At the end of the second stage, 7 or more patients out of the 17 enrolled should have survived with the native liver at 24 weeks post HMB002 treatment, to show evidence of efficacy of this novel hepatocyte transplantation that would support a larger randomised controlled trial.

Following signed informed consent from parent/legal guardian, the following screening tests and procedures will be undertaken to ensure patient is eligible to take part in the study (some of these may be part of routine care).

* Medical and Medication History
* Physical examination
* Height and weight monitoring
* Vital signs (body temperature, blood pressure, Pulse rate and Oxygen saturation)
* Urine or serum pregnancy test in females of childbearing potential
* Clinical blood tests and additional research bloods
* Recording of neurological parameters
* Ultrasound of the abdomen
* Quality of Life - Parent and where appropriate patient questionnaires (optional)

Enrolled participants will have pre-infusion checks and monitoring in the paediatric high dependency unit (HDU) or Paediatric intensive care unit (PICU). Children with acute liver failure generally require this degree of monitoring in any case. The child may be intubated and ventilated as part of routine care. This involves ventilation using a machine to help move air into and out of the lungs. If a suitable donor liver becomes available within 12 hours of planned study treatment, patient will go onto receive a liver transplant.

Following successful pre-infusion checks, the solution containing beads will be infused manually into the peritoneal cavity with usually a 50ml syringe, as a single infusion or several infusions, to achieve in excess of 25 million hepatocytes per kilogram of the body weight. HMB002 infusion will be done under ultrasound guidance.

* Participants will be continuously monitored before and for at least 24 hours after infusion in PICU/HDU. Some of these tests outlined below will be as per HDU and PICU standard of care. Once clinical condition permits and after 24 hours post infusion, the child may be stepped down to the paediatric wards.

  * Physical and neurological examination
  * Intra-abdominal pressure will be measured using urinary catheter where possible, at regular intervals both before and after infusion.
  * Regular review of the IMP infusion site
  * regular Vital signs (body temperature, blood pressure, Pulse rate and Oxygen saturation) • Clinical bloods at regular intervals both pre and post infusion.
  * Additional research bloods
  * Recording of ventilator settings and additional supportive therapy given as part of standard of care • Ultrasound of the abdomen
  * Recording of side effects
  * Recording of change in medications
* Participants will undergo daily examination until Day 7 while still an inpatient, and then be followed up at weeks 2, 4, 8, 12, 16, 24 and 52. Participants will be discharged following a liver organ transplant or upon recovery of their native liver. Therefore some of the follow up visits will be done in the outpatient clinics at King's College Hospital. Patients will have some or all of the assessments below at each follow up visit. Some of these visits will be part of standard routine care.

  * Physical and neurological examination
  * Height and weight monitoring,
  * Monitoring of Vital signs (body temperature, blood pressure, Pulse rate and Oxygen saturation)
  * Clinical Blood tests and additional bloods for research (at some visits; optional)
  * Recording of level of ventilator settings and supportive treatment as given with routine care.
  * Recording of side effects
  * Recording of changes to Medication
  * Parent and where appropriate patient questionnaires at final visit (optional parents/legal guardian consent
  * Ultrasound of the abdomen at specified time points in the protocol.

Microbeads will ideally be removed within 4 weeks of infusion. This will be done at the time of liver transplant or upon recovery of the native liver prior to discharge (using laparoscopy, a small key hole surgery of the abdomen).

Participants will also be followed up for another 9 years after HMB0002 infusion for monitoring of long term safety. This will be aligned with routine care and will be conducted annually as a minimum but may be more frequent depending on the clinical condition of the child or young person. Clinical blood tests and abdominal ultrasound data will be collected annually during the long term follow up period (years 2 to 5 as per routine care). SAEs (with exceptions) will be collected for the duration of the follow up period as outlined in the study protocol.

ELIGIBILITY:
Inclusion Criteria:

* Infant or child (male or female) under the age of 16 years at recruitment.
* Written informed consent obtained from a parent / legal guardian
* Presence of ALF defined as a multisystemic disorder in which severe impairment of liver function with or without encephalopathy occurs in association with hepatocellular necrosis reflected as synthetic liver failure in a child with no recognised underlying chronic liver disease. Children must fit one of the ALF categories as described in Appendix 1b(study protocol);
* Willing and able to comply with the study visit schedule.

Exclusion Criteria:

* Severe ascites causing high intra-abdominal pressure and / or respiratory compromise;
* Intra-abdominal sepsis suspected or proven;
* Clinical condition too unstable to tolerate procedure without compromise;
* Proven pre-existing allergy or intolerance to alginate on medical history;
* Proven pre-existing allergy to gentamicin on medical history;
* Intraperitoneal or intra-abdominal malignancy;
* Adhesions or fistulae to anterior abdominal wall;
* Children who weigh in excess of 33kg
* Pregnant or lactating patients (positive pregnancy test for females of child bearing potential at screening).
* Female patients of childbearing potential who are not willing to use highly effective methods of contraception to prevent pregnancy or abstain from heterosexual activity for 52 weeks post treatment.

  *Females of child bearing potential are females who have experienced menarche and are not surgically sterilised (e.g. by tubal occlusion, hysterectomy, bilateral salpingectomy) or post-menopausal (defined as at least 1 year since last regular menstrual period).

  ** Highly effective methods of birth control are those with a failure rate of < 1% per year when employed consistently and correctly. Highly effective methods of contraception as per HMA / CTFG working group are combined (Estrogen and Progestogen containing) hormonal contraception associated with inhibition of ovulation, the preparation may be oral, intravaginal or transdermal; progesterone-only hormonal contraception associated with inhibition of ovulation which may be oral, injectable or implantable; intrauterine device (IUD); intrauterine hormone-releasing system (IUS); bilateral tubal occlusion; vasectomised partner; sexual abstinence for 52 weeks post study treatment;

  *** Sexual abstinence is considered to be highly effective method only if defined as refraining from heterosexual activity from the date of consent until the week 52 visit post study treatment. The reliability of this method should be evaluated in relation to the duration of the study and the preferred and usual lifestyle of the participant.
* Male patients who are not willing to use an effective method of contraception (condom, vasectomy, sexual abstinence) for 52 weeks post study treatment, when engaging in sexual activity with a female of childbearing potential;
* Participation in concurrent therapeutic trial for ALF;
* Imminent liver transplantation expected within 12 hours of infusion;
* Total hepatectomy;
* Dependent on Extracorporeal Membrane Oxygenation (ECMO);
* Previous liver transplant

Max Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 17 (Estimated)
Dates: Start 2022-09 (Estimated); Primary Completion 2025-11 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Safety: Moderate to severe (including life threatening and death) adverse event occurrences due to product in 1st 52 weeks post procedure | Baseline to 52 weeks
  As above
Tolerability: assessed by the proportion of initiated infusion where >80% of the infusion is received by the patient. | 1 Day
  Tolerability: assessed by the proportion of initiated infusion defined by >80% of the IMP infusion is received by the patient on Day 0.
Biological activity: Survival with native liver at 24 weeks post treatment. | baseline to 24 weeks
  As above

SECONDARY OUTCOMES:
Change in blood marker levels including haematological, biochemical and coagulation baseline to 52 weeks post treatment. | Baseline to 52 weeks
  Change in full blood count and differentials, INR, APTT, fibrinogen, Serum levels of ALT, AST, Creatine Kinase, Total bilirubin, Conjugated bilirubin, Alkaline phosphatase, Albumin, total protein, serum urea, serum levels of sodium, potassium, chloride, urea, creatinine and plasma Ammonia - from baseline to 52 weeks post treatment.
Change in Quality of life measures from baseline to week 52 | Baseline and 52 weeks
  PedsQLTM Quality of Life Inventory questionnaires for parent and child will be completed at screening and week 52 visits. PedsQL - Parent Report for Infants, PedsQL - Parent Report for Toddlers (ages 2-4), PedsQL - Parent Report for Young Children (ages 5-7), PedsQL - Young Child Report (ages 5-7), PedsQL - Parent Report for Children (ages 8-12), PedsQL - Child Report (ages 8-12), PedsQL - Parent Report for Teenagers (ages 13-18), PedsQL - Teenager Report (ages 13-18) will be used. The items will be scored as per instructions on https://www.pedsql.org/score.html
Patient survival with native liver at 52 weeks post treatment | Baseline to 52 weeks
  As above
Patient survival with transplanted or native liver at 24 and 52 weeks post treatment. | Baseline to 24weeks and then 52 weeks
  As above

OTHER OUTCOMES:
To compare the ratios of specific SNP combinations in proteins between patients and donor cells by targeted mass spectrometry to distinguish the patient and recepient derived proteins | Baseline to 52 weeks
  As above
To analyse viability using fluorescent stains and function through the measurement of albumin of hepatocytes in microbeads which are retrieved from the intraperitoneal cavity either at laparoscopy or transplant for phenotype ex vivo. | Anytime within the 52 week period following investigational ,medicinal product infusiomn
  To evaluate the the hepatocytes in microbeads for viability of using fluorescent stains and cell function through the measurement of albumin

CONTACTS AND LOCATIONS:
Overall Officials: Anil Dhawan, Professor, Principal Investigator — King's College Hospital NHS Trust

IPD SHARING:
Plan to Share IPD: No
No plan to share identifiable patient data with other researchers.